CLINICAL TRIAL: NCT07096648
Title: Alert Burden When Monitoring Patients at Home
Acronym: WARD-HOME I
Status: Active, not recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Emilie Sigvardt, MD, Bispebjerg Hospital
Other Study IDs: H-20009132/91724
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Continuous Monitoring; Vital Signs Monitoring; Hospital at Home; Remote Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients discharged from hospital after admission due to an acute medical condition
  Interventions: Device: Continuous vital sign monitoring

INTERVENTIONS:
Device: Continuous vital sign monitoring — Continuous monitoring of vital signs performed using up to three CE- and FDA approved devices measuring heart rate, respiratory rate, systolic- and diastolic blood pressure, and SpO2. Data is transmitted to a CE-approved smartphone application that generates alerts in response to deviations based on predefined thresholds for duration and severity.

SUMMARY:
The aim of this observational study is to evaluate the burden and clinical relevance of vital sign alerts during home monitoring in recently discharged medical patients.

The primary outcome is the total number of vital sign alerts per patient per day. Secondary outcomes include the number of alerts per specific vital sign parameter, the frequency of alerts during daytime versus evening and nighttime, and the peak alert time during the day.

We will compare alert data without filtering to data processed with AI-driven filtering methods to assess if these filters reduce the number of non-actionable alerts while maintaining clinical relevance.

Participants will be equipped with wearable devices to continuously monitor heart rate, respiratory rate, blood pressure, and oxygen saturation during the first days after hospital discharge. Vital signs will be transmitted remotely, and alerts will be generated based on predefined thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted with an acute medical disease and scheduled for discharge within five days from inclusion.

Exclusion Criteria:

* Allergy to plaster/silicone, pacemaker or ICD, inability to give informed consent or deemed not able to open the front door when visited by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from Copenhagen University Hospital - Bispebjerg and Frederikberg. Eligible patients are enrolled in the study at the time of hospital discharge following admission for an acute medical condition.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of vital sign alerts per patient per day | Up to 8 days

SECONDARY OUTCOMES:
Number of alerts per specific vital sign parameter per patient per 24-hour period | Up to 8 days
Frequency of any vital sign alert per hour analyzed as daytime (08.00-15.59) vs. evening and nighttime (16.00-07.59) | Up to 8 days
The hour of day with highest frequency of alerts | up to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, Professor, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark